CLINICAL TRIAL: NCT07188805
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Phase 3 Study to Investigate the Efficacy, Safety, and PK/ PD of Finerenone, in Addition to Standard-of-care, in Pediatric Patients, 6 Months to < 18 Years of Age With Heart Failure (HF) and Left Ventricular Systolic Dysfunction (LVSD)
Brief Title: A Study to Learn More About How Well Finerenone Works, How Safe it is, and How it Moves Into, Through, and Out of the Body Compared to Placebo When Taken With Standard Treatment in Children With Heart Failure and Left Ventricular Systolic Dysfunction
Acronym: FIORE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 21466; 2024-519829-38-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2025-09-08; First posted 2025-09-23 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Left Ventricular Systolic Dysfunction; Heart Failure (Pediatric)
MeSH Terms: conditions — Ventricular Dysfunction, Left; Heart Failure | interventions — finerenone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Finerenone (Kerendia, BAY94-8862) (Experimental): Participants will receive finerenone treatment.
  Interventions: Drug: Finerenone (Kerendia, BAY94-8862)
- Placebo (Placebo Comparator): Participants will receive placebo to finerenone.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Finerenone (Kerendia, BAY94-8862) — Finerenone in different doses, treatment duration will be 90±3 days
  Arms: Finerenone (Kerendia, BAY94-8862)
Drug: Placebo — Placebo to finerenone, treatment duration will be 90±3 days
  Arms: Placebo

SUMMARY:
Researchers are looking for a better way to treat children who have heart failure with left ventricular systolic dysfunction (LVSD). Heart failure is a serious condition where the heart is unable to pump enough blood to meet the body's needs. This can lead to symptoms like shortness of breath, fatigue, and poor growth in children.

The study treatment, finerenone (also called BAY94-8862), works by blocking a protein involved in inflammation, scarring, and thickening of the heart and blood vessels. This may help the heart to pump blood more effectively. This is the first study to explore its use specifically for children with heart failure and LVSD.

The main purpose of this study is to learn if finerenone works to help the heart compared to placebo in children with heart failure and LVSD. For this, the researchers will collect and analyze data on the levels of a protein called NT-proBNP in the blood, which indicates heart stress, and monitor the safety of the treatment.

The study will include children with heart failure and LVSD aged from 6 months to less than 18 years. The study participants will be randomly assigned to one of two treatment groups. Based on their group, they will receive either finerenone or a placebo for a duration of 3 months. A placebo looks like a treatment but does not have any medicine in it. Throughout the study, all participants will continue to receive their standard heart failure treatments.

At the start of this study, the doctors will check each participant's medical history and current medications. If participants qualify for the treatment phase, they will undergo treatment for about 90 days. During this time, they will visit the study site at least 3 times. During these visits, the participants will:

* have their blood pressure, heart rate, temperature, respiratory rate, height and weight measured
* have their heart examined by electrocardiogram (ECG) and echocardiogram
* have blood samples taken
* have physical examinations
* answer questions about their medication and whether they have any adverse events, or have their parents or guardians' answers

An adverse event is any medical problem that a participant has during a study. Doctors keep track of all adverse events that happen in studies, even if they do not think the adverse events might be related to the study treatments.

After the initial three-month study, eligible participants will have the option to join a nine-month open-label extension study where all will receive finerenone. Participants who choose not to enroll in the extension will have a follow-up visit 30 days after their last treatment.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 6 months to <18 years old at the time when the informed consent/assent is signed.
* Left ventricular systolic dysfunction (LVSD) with left ventricular ejection fraction (LVEF) ≤ 50% at screening assessed by echocardiography.
* Elevated NT-pro BNP levels

  * >500 ng/l for children ≥ 6 months to < 2 years of age
  * >300 ng/l, for children ≥ 2 years to <18 years
* Heart failure etiologies including congenital heart defects (CHD) with biventricular physiology and systemic LV; idiopathic cardiomyopathy (CM); familial/inherited and/or genetic CM; history of myocarditis (diagnosis of an acute episode was at least 3 months prior to randomization); neuromuscular disorder (eg, duchenne muscular dystrophy); inborn error of metabolism; mitochondrial disorder; acquired (chemotherapy, iatrogenic, infection, rheumatic, or nutritional); ischemic (eg, Kawasaki disease and postoperative heart failure [HF]); LV noncompaction.
* Receiving standard of care (SoC) treatment for heart failure according to local guidelines or investigator´s discretion and being on a stable regimen for 30 days prior to randomization.
* Study participants must have a body weight ≥ 4.0 kg at Visit 1.

Exclusion Criteria:

* Serum potassium:

  * > 5.0 mmol/L for children ≥ 2 years of age at either screening or randomization visit
  * > 5.3 mmol/L for children ≥ 6 months to < 2 years of age at either screening or randomization visit (if estimated glomerular filtration rate [eGFR] < 60 mL/min/1.73m², threshold of > 5.0 mmol/L will be used)
* Severe renal dysfunction with eGFR < 30 ml/min/1.73m² at screening or randomization visit.
* Systolic blood pressure (SBP) < 5th percentile for age, sex and height at screening or randomization.
* Sustained or symptomatic arrhythmias not controlled by drug or device therapy within 30 days prior to randomization.
* Treatment with a mineralocorticoid receptor antagonist (e.g., spironolactone, eplerenone) within 30 days of randomization.
* Requirement of any intravenous (IV) vasoactive agents, mechanical ventilation, mechanical circulatory support within 30 days prior to randomization.
* Recent surgical procedure or other intervention to correct or palliate CHD within 3 months prior to randomization or anticipated to undergo cardiac surgery during the 3 months after randomization.

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 111 (Estimated)
Dates: Start 2025-11-19 (Actual); Primary Completion 2029-11-30 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in NT-proBNP levels | From baseline to Day 90±3

SECONDARY OUTCOMES:
Number of participants with treatment-emergent adverse events (TEAEs) | From the start of study intervention to last study intervention (up to 93 days) + 3 days
  TEAEs will be mapped to Medical Dictionary for Regulatory Activities (MedDRA) terms
Change in serum potassium levels | From baseline to Day 90±3
Change in estimated glomerular filtration rate (eGFR) | From baseline to Day 90±3
Change in systolic blood pressure (SBP) | From baseline to Day 90±3
Change in left ventricular systolic function | From baseline to Day 90±3
  Change measured by echocardiogram (%) from baseline to Day 90±3
Total number of cardiovascular outcome events, including cardiovascular death, heart transplantation, and clinical worsening of heart failure | From baseline to Day 90±3
Maximum observed finerenone concentration in plasma after multiple doses (Cmax, md) | Pre-dose, post-dose (1.5-5 hours after intake of intervention), up to day 90±3
Area under the curve for finerenone concentration in plasma after multiple doses (AUCτ,md) | Pre-dose, post-dose (1.5-5 hours after intake of intervention), up to day 90±3

CONTACTS AND LOCATIONS:
Locations (133):
- United States (22):
  - Children's Hospital Colorado - Anschutz Medical Campus - Cardiology, Aurora, Colorado
  - Nemours Children's Hospital - Delaware - Cardiology, Wilmington, Delaware
  - UF Health Shands Hospital - Pediatric Cardiology, Gainesville, Florida
  - Joe Dimaggio Children's Hospital - Cardiology, Hollywood, Florida
  - Emory University Hospital - Children's Healthcare of Atlanta Cardiology - Atlanta, Atlanta, Georgia
  - Riley Hospital For Children - Cardiology, Indianapolis, Indiana
  - Boston Children's Hospital - Main Campus - Cardiology, Boston, Massachusetts
  - C.S. Mott Children's Hospital - Cardiology, Ann Arbor, Michigan
  - Children's Mercy Hospital Kansas City - Cardiology, Kansas City, Missouri
  - Washington University - St. Louis Children's Hospital - Cardiology, St Louis, Missouri
  - Icahn School of Medicine at Mount Sinai - Pediatric Cardiology, New York, New York
  - Columbia University Irving Medical Center - Pediatric Cardiology, New York, New York
  - The Children's Hospital at Montefiore - Cardiology, The Bronx, New York
  - Cincinnati Children's Hospital Medical Center | Division of Nephrology and Hypertension, Cincinnati, Ohio
  - Cleveland Clinic Children's, Cleveland, Ohio
  - Nationwide Children's Hospital - Cardiology, Columbus, Ohio
  - Children's Hospital of Philadelphia - Cardiology, Philadelphia, Pennsylvania
  - UPMC Children's Hospital of Pittsburgh - Cardiology, Pittsburgh, Pennsylvania
  - MUSC Shawn Jenkins Children's Hospital - Cardiology, North Charleston, South Carolina
  - Children's Medical Center Dallas - Cardiology, Dallas, Texas
  - Texas Children's Hospital - Cardiology, Houston, Texas
  - Eccles Primary Children's Outpatient Services - Cardiology, Salt Lake City, Utah
- Argentina (10):
  - Hospital de Niños Sor María Ludovica, La Plata, Buenos Aires
  - Instituto De Investigaciones Clinicas Zarate | Zarate, Argentina, Zárate, Buenos Aires
  - Hospital General de Ninos Ricardo Gutierrez | Pediatric Nephrology Department, Buenos Aires, Ciudad Auton. de Buenos Aires
  - Consultorios Integrados Rosario | Instituto Medico de la Fundacion de Estudios Clinicos, Rosario, Santa Fe Province
  - Hospital Italiano de Buenos Aires, Buenos Aires
  - Hospital de Pediatría Juan P. Garrahan, Buenos Aires
  - Hospital General de Ninos Pedro de Elizalde | Nephrology Department, Ciudad Autonoma de Buenos Aire
  - Consultorios Médicos Dr. Doreski, Ciudad Autónoma de Buenos Aire
  - Sanatorio de la Cañada, Córdoba
  - Centro Cardiovascular Salta (Torzav SRL), Salta
- Austria (2):
  - Kepler Universitätsklinikum GmbH - Klinik für Kinderkardiologie, Innsbruck, Upper Austria
  - Medizinische Universität Wien - Klinik für Kinder- und Jugendheilkunde, Abteilung für Pädiatrische Kardiologie, Vienna, Vienna
- Belgium (5):
  - UZ Leuven - Pediatric Cardiology, Leuven, Flemish Brabant
  - Cliniques Universitaires St-Luc (UCL) - Pediatric Cardiology, Brussels
  - UZ Antwerpen - Pediatric Cardiology, Edegem
  - UZ Gent - Pediatric Cardiology, Ghent
  - CHC MontLegia - Pediatric Cardiology, Liège
- Brazil (10):
  - Instituto Dante Pazzanese de Cardiologia | Divisao de Pesquisa, São Paulo, Ceará
  - InCor HCFMUSP, São Paulo, Ceará
  - Hospital de Clínicas da Universidade Federal de Uberlândia Empresa Brasileira de Serviços Hospitalares - EBSERH, Uberlandia, Espírito Santo
  - Hospital Pequeno Principe, Curitiba, Estado de Bahia
  - Hospital Infantil Sabará - Instituto PENSI - Pesquisa e Ensino em Saúde Infantil, São Paulo, Minas Gerais
  - IESG - Instituto de Ensino da Saude e Gestao, São Paulo, Rio Grande do Norte
  - Santa Casa de Misericórdia de Belo Horizonte, São Paulo, Rio Grande do Sul
  - Fundação Universidade de Caxias do Sul, Marília, São Paulo
  - Centro de Pesquisa Clinica e Populacional Hospitalize, Porto Alegre, São Paulo
  - Campinas Clinical Research Institute (IPECC) | Campinas, Brazil, São Paulo, São Paulo
- Bulgaria (4):
  - National Heart Hospital (NHH) - Dept. Pediatric Cardiology, Sofia, Sofia
  - University Multiprofile Hospital for Active Treatment 'Sveti Georgi' EAD, Plovdiv Pediatric Clinic, Plovdiv
  - Medical Center Nora- Heart ?OOD Child Cardiology, Sofia
  - University Multiprofile Hospital for Active Treatment 'Sveta Ekaterina' EAD, Sofia, Sofia
- Canada (6):
  - Stollery Children's Hospital (SCH), Edmonton, Alberta
  - BC Children's Hospital - Children's Heart Centre, Vancouver, British Columbia
  - London Health Sciences Centre - Children's Hospital, London, Ontario
  - The Hospital for Sick Children (SickKids), Toronto, Ontario
  - CHU Sainte-Justine, Montreal, Quebec
  - University of Saskatchewan, Royal University Hospital, Saskatoon, Saskatchewan
- Czechia (2):
  - Fakultní nemocnice Brno, Detská nemocnice - Pediatrická klinika, Brno
  - Fakultní nemocnice Motol a Homolka, Pracovište MOTOL - Detské kardiocentrum 2. LF UK a FN Motol, Prague
- Finland (2):
  - HUS-Yhtymä, Helsingin yliopistollinen sairaala (HUS) - Uusi lastensairaala, kardiologia, Helsinki
  - Oulu University Hospital, Oulun yliopistollinen sairaala (OYS) - Lasten ja nuorten palvelut, Oulu
- Germany (3):
  - Universitaetsklinikum Giessen und Marburg GmbH - Kinderherzzentrum und Zentrum für angeborene Herzfehler, Giessen, Hesse
  - Universitätsklinikum Köln - Kinderkardiologie, Cologne
  - Universitätsklinikum Tübingen, Kinderheilkunde II - Kinderkardiologie, Pulmologie, Intensivmedizin, Tübingen
- Greece (4):
  - Onassis Cardiac Surgery Center, Department of Pediatric Cardiology and Adult Congenital Heart Disease, Kallithea, Attica
  - Athens General Children's Hospital Panagioti And Aglaia Kyriakou -2nd University Department of Pediatrics, Athens
  - Athens General Children's Hospital Panagioti And Aglaia Kyriakou, Cardiology Department, Athens
  - Nosokomeio Paidon I Agia Sofia, Cardiology Department, Athens
- Gottsegen Gyorgy Orszagos Kardiovaszkularis Intezet - Gyermeksziv Kozpont, Budapest, Hungary
- Israel (5):
  - Rambam Health Corporation, Haifa
  - Edith Wolfson Medical Center (EWMC), Holon
  - Shaare Zedek Medical Center, Jerusalem
  - Dana-Dwek Children's Hospital, Tel Aviv
  - Chaim Sheba Medical Center, Tel Litwinsky
- Italy (8):
  - Azienda Socio Sanitaria Territoriale Papa Giovanni XXIII - Cardiologia 2 - Cardiopatie Congenite del bambino e dell'adulto, Bergamo
  - Azienda Ospedaliero-Universitaria di Bologna IRCCS Policlinico Sant'Orsola-Cardiologia pediatrica ed dell'età evolutiva, Bologna
  - IRCCS Istituto Giannina Gaslini - Cardiologia, Genova
  - ASST Grande Ospedale Metropolitano Niguarda - Struttura semplice dipartimentale cardiologia pediatrica, Milan
  - Azienda Ospedaliera Dei Colli_Monaldi - Malattie Rare e Genetiche Cardiovascolari, Naples
  - Azienda Ospedale-Università di Padova - UOC Cardiologia Pediatrica, Padua
  - Ospedale Pediatrico Bambino Gesù - Unità Terapie Cardiovascolari Avanzate, Roma
  - A.O.U. Città della Salute e della Scienza di Torino_Regina Margherita - Cadiologia pediatrica, Torino
- Mexico (8):
  - Centro de Investigación Clínica Médica y Farmacológica S.A de C.V, Guadalajara, Jalisco
  - Hospital Infantil de México "Dr. Federico Gómez", Mexico City, Mexico City
  - Hospital Universitario "Dr. Jose Eleuterio Gonzalez"-Pediatria, Monterrey, Nuevo León
  - Invecordis Sc., Huixquilucan, State of Mexico
  - Centro de Estudios de Investigacion Metabolicos y Cardiovasculares, Ciudad Madero, Tamaulipas
  - Centro de Estudios Clínicos de Querétaro S.C., Querétaro
  - Centro de Atención e Investigación Cardiovascular del Potosí S.C., San Luis Potosí City
  - Instituto Nacional de Cardiología "Ignacio Chávez", Tlalpan
- Poland (4):
  - Wojewodzki Szpital Specjalistyczny we Wroclawiu, Wroclaw, Lower Silesian Voivodeship
  - Pomnik Centrum Zdrowia Dziecka - Klinika Kardiologii, Warsaw, Masovian Voivodeship
  - Górnoslaskie Centrum Zdrowia Dziecka im. sw. Jana Pawla II SPSK Nr 6 Slaskiego UM w Katowicach - Oddzial Kardiologii Dzieciecej, Katowice
  - Instytut Centrum Zdrowia Matki Polki w Lodzi - Klinika Kardiologii, Lódz
- Portugal (5):
  - Hospital de Santa Cruz | Pediatric Cardiology Department, Carnaxide
  - Department of Cardiology - Research Unit, Coimbra
  - Hospital Santa Marta | Pediatric Cardiology Department, Lisbon
  - Centro Materno infantil do Norte - Pediatric Cardiology, Porto
  - ULS São João - Pediatric Department, Porto
- South Korea (4):
  - Pusan National University Yangsan Children's Hospital, Yangsan, Gyeongsangnam-do
  - Seoul National University Hospital-Pediatrics Department, Jongno, Seoul
  - Severance Hospital, Yonsei University Health System-Pediatrics Department, Seodaemun
  - Samsung Medical Center-Pediatrics, Seoul
- Spain (8):
  - Hospital Sant Joan De Deu Barcelona | Cardiologia pediatrica, Esplugues de Llobregat, Barcelona
  - Hospital Universitari Vall D Hebron | Cardiologia pediatrica, Barcelona
  - Hospital Universitario Reina Sofia | Cardiologia pediatrica, Córdoba
  - Hospital Universitario Ramon Y Cajal | Cardiologia pediatrica, Madrid
  - Hospital Universitario 12 De Octubre | Cardiologia pediatrica, Madrid
  - Hospital Universitario La Paz | Cardiologia pediatrica, Madrid
  - Hospital Universitario Regional De Malaga | Cardiologia pediatrica, Málaga
  - Hospital Universitario Virgen Del Rocio S.L. | Cardiologia pediatrica, Seville
- Skånes Universitetssjukhus Lund - Barnhjärtcentrum, Lund, Skåne County, Sweden
- Taiwan (6):
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - Chang Gung Memorial Hospital Kaohsiung, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - MacKay Children's hospital, Taipei
- Turkey (Türkiye) (6):
  - Cukurova Universitesi Tip Fakultesi Hastanesi, Adana
  - Hacettepe Universitesi Tip Fakultesi, Ankara
  - Ankara Bilkent Sehir Hastanesi, Bilkent Ankara
  - Marmara Uni. Tip Fak. Pendik EAH Kardiyoloji, Istanbul
  - Istanbul Mehmet Akif Ersoy Gogus Kalp Damar Cerrahisi E.A.H., Istanbul
  - Izmir Dr. Behcet Uz Cocuk Hastaliklari Hast, Izmir
- United Kingdom (7):
  - University Hospitals of Leicester NHS Trust | Leicester Children's Hospital - Children's Research Facility, Leicester, Leicestershire
  - Alder Hey Children's NHS Foundation Trust | Alder Hey Children's Hospital - Clinical Research Facility, Liverpool, Merseyside
  - Belfast Health and Social Care Trust | Royal Belfast Hospital for Sick Children - Paediatric Cardiology, Belfast, Northern Ireland
  - NHS Greater Glasgow and Clyde | Royal Hospital for Children - Glasgow Clinical Research Facility, Glasgow, Scotland
  - Newcastle upon Tyne Hospitals NHS Foundation Trust |Freeman Hospital - Children's Heart Unit, Newcastle upon Tyne, Tyne and Wear
  - Leeds Teaching Hospitals NHS Trust | Leeds Children's Hospital - Children's Research Facility, Leeds, West Yorkshire
  - University Hospitals Bristol and Weston NHS Foundation Trust | Bristol Royal Hospital for Children - Clinical Research Facility, Bristol

IPD SHARING:
Plan to Share IPD: No
Currently, there is no established plan for the sharing of Individual Patient Data (IPD) from this study. The availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA 'Principles for responsible clinical trial data sharing.' This pertains to the scope, timepoint, and process of data access.
  As such, Bayer commits to considering requests from qualified researchers for patient- / study-level clinical trial data, and documents from clinical trials involving medicines and indications approved in the US and EU. However, this commitment does not reflect an active IPD sharing plan. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Researchers can use www.vivli.org to request access to IPD and documents from clinical studies to conduct research. Information on Bayer's criteria for listing studies is provided in the member section of the portal.

REFERENCES:
- See also: Click here to find further information and, after study completion, the study results according to Bayer's transparency standards. — https://clinicaltrials.bayer.com/study/21466